CLINICAL TRIAL: NCT01887431
Title: Telecare in Adults With Type 1 Diabetes Mellitus Treated by Insulin Pump - A Randomized Controlled Trial
Brief Title: Telecare in Type 1 Diabetes (T1D) Patients Treated by Insulin Pump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Principal Investigator, Bruria Sher, Dietitian, Assuta Hospital Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 71156
Record Dates: First submitted 2013-06-18; First posted 2013-06-26 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes Mellitus, Type 1; Adult; Insulin Infusion Systems; Telecare
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telecare (Experimental): Each patient will transmit glucometer and pump data electronically via a web site to diabetes team and will receive feedback by telephone. Frequency of data transfer will be directly related to patients' metabolic control.
  Interventions: Other: Telecare
- Conventional therapy (Active Comparator): 3-month routine clinic visits
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: Telecare — Each patient will transmit glucometer and pump data electronically via a web site (Medtronic Carelink internet site www.carelink.minimed.com) to diabetes team and will receive feedback by telephone. Frequency of data transfer will be directly related to patients' metabolic control. In addition to data transmission Patient of the intervention group will be arriving during the intervention year for 3 clinic visit at the following time point : 0, 6 and 12 month.
  Arms: Telecare
Other: Conventional therapy — 3-month routine clinic visits
  Arms: Conventional therapy

SUMMARY:
The purpose of this study is to determine whether Telecare can be used for efficient management of adults with Type 1 Diabetes Mellitus using insulin pump, in lieu of frequent clinic visits.

DETAILED DESCRIPTION:
1. Objectives

   1. To evaluate the effect of telecare on glycemic control for patients with type 1 diabetes (T1DM).
   2. To assess the cost of telecare to Maccabi, the patient and the economy.
   3. To assess patients' quality of life and satisfaction with telecare intervention.
   4. To assess the effect of telecare intervention on insulin adjustment to consumed carbohydrates.
2. Working hypothesis Telecare can be used for efficient management of T1DM in adults using insulin pump, in lieu of frequent clinic visits.
3. Methodology A randomized controlled prospective trial for one year. Intervention group: Each patient will transmit glucometer and pump data electronically via a web site (Medtronic Carelink internet site www.carelink.minimed.com) to diabetes team and will receive feedback by telephone. Frequency of data transfer will be directly related to patients' metabolic control. In addition to data transmission Patient of the intervention group will be arriving during the intervention year for 3 clinic visit at the following time point : 0, 6 and 12 month.

   Control group: 3-month routine clinic visits
4. Significance of the proposed research (its uniqueness and innovation) Telecare potentially offers a method for efficient continuous care management of patients with T1DM using insulin pump in lieu of clinic visits. It enables real time responses of clinical personnel and increases patient involvement. This trial will be the first telecare intervention lasting for one year to determine if treatment is as efficient as face to face visits, thus enabling cost reduction and time saving without affecting the quality of care. .

ELIGIBILITY:
Inclusion Criteria:

* Patients with T1D lasted >1 year, age 22 and up, using insulin pump
* Patients possessing a mobile phone and internet access

Exclusion Criteria:

* Patients with Severe target organ damage
* Patients with Mental retardation
* Patients with Eating disorders
* Pregnant patients or patients planning pregnancy

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated Hemoglobin (Hba1c) | From date of randomization every 3 months, up to one year

SECONDARY OUTCOMES:
Time spent on data analysis and telephone calls by team | 1 year
Number of severe hypoglycemic and diabetic ketoacidosis (DKA) events and hospitalizations | 1 year
Patients' quality of life | 1 year
Patients' satisfaction | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Maccabi Healthcare Services, Raanana, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yaron M, Sher B, Sorek D, Shomer M, Levek N, Schiller T, Gaspar M, Frumkin Ben-David R, Mazor-Aronovitch K, Tish E, Shapira Y, Pinhas-Hamiel O. A randomized controlled trial comparing a telemedicine therapeutic intervention with routine care in adults with type 1 diabetes mellitus treated by insulin pumps. Acta Diabetol. 2019 Jun;56(6):667-673. doi: 10.1007/s00592-019-01300-1. Epub 2019 Feb 19. PMID 30783823